CLINICAL TRIAL: NCT02825446
Title: A Pilot Prospective Study of Two Methods of Revascularization of Tibial Arteries: Angioplasty Tibial Arteries, and Angioplasty Tibial Artery, Augmented by Radio Frequency Denervation Popliteal Artery in Patients With Steno-occlusive Lesion of the Tibial Arteries
Brief Title: Angioplasty of the Tibial Arteries Augmented Radio Frequency Denervation of the Popliteal Artery
Acronym: ATRFPA
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: a significant number of patients were not selected
Sponsor: Meshalkin Research Institute of Pathology of Circulation (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: N-RICP-873
Record Dates: First submitted 2016-06-28; First posted 2016-07-07 (Estimated); Last update posted 2020-07-08 (Actual); Status verified 2020-05

CONDITIONS: Сhronic Ischemia of the Lower Extremities; Atherosclerosis of the Tibial Arteries; Lesion no More Than Two Tibial Arteries; Steno-occlusive Lesion of the Tibial Arteries
Keywords: radio frequency denervation; tibial arteries; atherosclerosis of the peripheral arteries

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- angioplasty tibial arteries (Active Comparator)
  Interventions: Procedure: angioplasty tibial arteries
- radio frequency denervation popliteal artery by the use (Experimental): radio frequency denervation popliteal artery "Vessix Renal Denervation System Balloon"
  Interventions: Procedure: angioplasty tibial arteries augmented radio frequency denervation popliteal artery by the use"Vessix Renal Denervation System Balloon"

INTERVENTIONS:
Procedure: angioplasty tibial arteries — Under local anesthesia using the standard endovascular access and renders the affected arterial segment. Are stenosis or occlusion of the artery, the hydrophilic guide. Occlusion or subintimal perform transluminal recanalization of the artery. Then do balloon angioplastic stenosis or occlusion.
  Drug therapy includes the administration of aspirin before the procedure (160-300 mg/day) starting at least one day, and heparin during the procedure (5000 IU intravenously). After the procedure, all patients are administered aspirin (100 mg daily) for a long time.
  Arms: angioplasty tibial arteries
Procedure: angioplasty tibial arteries augmented radio frequency denervation popliteal artery by the use"Vessix Renal Denervation System Balloon" — Under local anesthesia using the standard endovascular access and renders the affected arterial segment. Are stenosis or occlusion of the artery, the hydrophilic guide. Occlusion or subintimal perform transluminal recanalization of the artery. Then do balloon angioplastic stenosis or occlusion. Then in 3 portion of the popliteal artery starts ablation by the use "Vessix Renal Denervation System Balloon" performed radiofrequency denervation. After removal of the balloon, control angiography is performed.
  Drug therapy includes the administration of aspirin before the procedure (160-300 mg/day) starting at least one day, and heparin during the procedure (5000 IU intravenously). After the procedure, all patients are administered aspirin (100 mg daily) for a long time.
  Arms: radio frequency denervation popliteal artery by the use

SUMMARY:
Angioplasty augmented radiofrequency denervation popliteal artery, in our opinion, will remove the spasm with macro and microcirculatory blood flow, which increases revascularization patency of tibial arteries.

ELIGIBILITY:
Inclusion Criteria:

* Chronic lower limb ischemia 3-6 degree by Rutherford;
* Stenosis or occlusion of no more than 2 tibial arteries;
* Stenosis of the tibial arteries more than 70 %;
* Duration stenosis or occlusion no more than 70 mm;

Exclusion Criteria:

* Diabetes mellitus type 2
* Occlusion or stenosis of all tibial arteries
* Expressed calcification of tibial arteries angioplasty tolerant
* Hemodynamically significant stenosis of the popliteal artery;
* Chronic heart failure of III-IV functional class by NYHA classification;
* Decompensated chronic "pulmonary" heart;
* Severe hepatic or renal failure (bilirubin> 35 mmol / l, glomerular filtration rate <60 mL / min);
* Polyvalent drug allergy;
* Cancer in the terminal stage with a life expectancy less than 6 months;
* Patient refusal to participate or continue to participate in the study;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2020-06 (Actual)

PRIMARY OUTCOMES:
the absence of thrombosis or stenosis of the popliteal artery | 12 mounth after intervention
  during the whole period of observation, confirmation of patency of the arterial ultrasound of the operated segment as well as such parameters as flow rate, presence of stenosis (%) or thrombosis

SECONDARY OUTCOMES:
Primary patency after intervention | 12-mounth after intervention
  during the whole period of observation, confirmation of patency of the arterial ultrasound of the operated segment as well as such parameters as flow rate, presence of stenosis (%) or thrombosis
Secondary patency after intervention | 12-mounth after intervention
  during the whole period of observation, confirmation of patency of the arterial ultrasound of the operated segment as well as such parameters as flow rate, presence of stenosis (%) or thrombosis
Number of participants with limb salvage | 12 mounth after intervention
  Number of participants with limb salvage
Laser Doppler Flowmetry | 12 mounth after intervention
  to assess the microcirculation of the lower limbs use such parameters as:
  * the time until the maximal post-occlusive blood flow
  * maximal post-occlusive blood flow
  * post-occlusive blood flow increase of
Transcutaneous oxygen tension | 12 mounth after intervention
  to assess the microcirculation of the lower limbs use a level transcutaneous oxygen tension (%)

CONTACTS AND LOCATIONS:
Overall Officials: Andrey Karpenko, Study Director — Academician EN Meshalkin Novosibirsk State Budget Research Institute of Circulation Pathology
Locations (1):
- NRICP, Novosibirsk, Russia